CLINICAL TRIAL: NCT03596853
Title: Effects of the Addition of a Protocol of Progressive Mobilization With Dose Control and Training Load in in Critically Ill Patients: Randomized Controlled Trial
Brief Title: Progressive Mobilization With Dose Control and Training Load in in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Principal Investigator, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUBahia Mobilization ICU
Record Dates: First submitted 2018-06-21; First posted 2018-07-24 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking: Triple (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Mobilization (Experimental): These patients will receive standard rehabilitation delivered by non-study physiotherapist. In addition, the patients will undergo a protocol of progressive mobilization with individualized dose control and training load stratified according to functional levels and performance.
  Interventions: Other: Progressive mobilization
- Control: Usual care (Sham Comparator): These patients will receive standard rehabilitation delivered by non-study physiotherapist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Progressive mobilization — Will be applied once a day, 5x/ week, performed into 4 levels: N1 (bridge and rolling for both sides); N2 (transfer training from lying down to sitting on both sides); N3 (sit and stand up from a chair); N4 (running training). According to their functional level, patients will perform, once a day, 8 sets of each movement, alternating 20 seconds of execution with 10 seconds of rest. Patients will be stimulated constantly to perform the movements with the highest possible speed.
  If the patient performs adequately within of your level functional level, can will progress in level, if can not progress, there will be an increase in training volume within the level itself. Adequate performance within the functional level means that the patient is able to complete more than eight sets of exercise and does not present increased sensation of pain, present sensation of perceived exertion within the safety limit of the protocol (Borg ≤ 6).
  Arms: Experimental: Mobilization
Other: Usual Care — This group will receive standard usual, which will be monitored, but not protocolised.
  Arms: Control: Usual care

SUMMARY:
Immobilization and bed rest of patients in intensive care units (ICU) increases their risk for muscle dysfunction and prolonged mechanical ventilation, leading to physical deconditioning and loss of functionality. Active mobilization is a therapeutic strategy that typically involves exercises in which the patient uses his or her own strength and muscular control, is a feasible, safe, and low-cost intervention to improve muscle dysfunction and disability in patients at the ICU. Despite scientific advances, the current description and prescriptions of exercises at the ICU remain incomplete with respect to the control and the description of the variables of training load (volume and intensity), programming, and progression.

DETAILED DESCRIPTION:
This prospective double-blind (patient and evaluator). This study will be conducted in accordance with Consolidated Standards of Reporting Trials recommendations. The trial will be performed at the University Hospital Professor Edgard Santos in Salvador, Bahia, Brazil. This study was approved by the institutional hospital ethics committee (approval reference number 2.371.933). Before enrollment, written informed consent will be obtained from participants or their legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Being able to roll in the bed and bridge.
* Barthel score of at least 70 weeks before admission to the ICU
* Ability to interact with the researcher

Exclusion Criteria:

* Mortality rate in excess of 50% according to Acute Physiology and Chronic Health Disease Classification System II (APACHEII)
* Present intracranial pressure increase
* Cardiorespiratory arrest,
* Has unstable fractures that hamper progression in levels of mobilization,
* Severe lower limb injury or amputation
* Neuromuscular disease
* Underwent radiotherapy and / or chemotherapy in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Length of ICU stay in days | at 28 days or discharge from ICU whichever occurs earlier
  Time in days, from baseline to discharge from ICU

SECONDARY OUTCOMES:
Muscle mass | Change from baseline at 28th day
  Ultrasound measurement (quadriceps, biceps brachii, and diaphragm - cross-sectional area on B-mode ultrasound
Change in muscle strength | Baseline and after 3 and at 7 day intervals up to 28th day or discharge from ICU
  Muscle Strength measured by hand held dynamometer
Physical activity: total activity | At 28 days or discharge from hospital
  accelerometry measurement of the total activity
Activity and participation | Change from baseline up to 1 year post discharge
  Measurement characteristics of World Health Organisation Disability Assessment Schedule II
Mortality | At 28 days or discharge from hospital and at 12 months
  Mortality
Functional Status | Change from baseline up to 28th day or discharge from hospital
  Functional Status Measured Using Functional Status Score for the Intensive Care Unit (involves five functional tasks (rolling, supine to sit transfer, sit to stand transfer, sitting on the edge of bed and walking). Each task is evaluated using an 8-point ordinal scale ranging from 0 (not able to perform at all) to 7 (complete independence)
Surgical Optimal Mobilisation Score (SOMS) level | Change from baseline up to 28th day or discharge from hospital
  Surgical Optimal Mobilisation Score (SOMS) level algorithm for goal-directed mobility ranges from '0-No mobility' to '4-Ambulation'. The intermediate steps are '1-Passive Range of Motion,' '2-Sitting,' and '3-Standing.'
Mobility | Change from baseline up to 28th day or discharge from hospital
  Timed up-and-go score
Health-Related Quality of Life: SF-36 | At 28 days or discharge from hospital and at 12 months
  Health-Related Quality of Life will be measured by a questionnaire 36-item Short Form Health Survey. The SF-36 is a widely used generic instrument for evaluating HRQoL, consisting of eight subscales evaluating specific health status domains and two summary scales, a Physical Component Summary and a Mental Component Summary. Scores on the SF-36 range from 0 to 100, with higher scores indicating better health status.
Days with mechanical ventilation | From 3 to 28 days
  Number of uninterrupted days in use of mechanical ventilation
Length of hospital stay in days | Up to 1 month post hospital discharge
  Time in days, from baseline to discharge from hospital
Muscle thickness | Change from baseline at 28th day
  Ultrasound measurement (quadriceps, biceps brachii, and diaphragm on B-mode ultrasound measured in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Mansueto Gomes Neto, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided